CLINICAL TRIAL: NCT04957394
Title: Family Partner -Co-development, Implementation and Evaluation of a Child Maltreatment Prevention Intervention
Brief Title: Pilot Trial of Family Partner - a Child Maltreatment Prevention Intervention
Acronym: FAMPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: SOS Children's Villages, Norway (Unknown); Øvre Eiker municipality (Unknown); Lillehammer municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 804402
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Family; Parenting; Child Maltreatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Family Partner) (Experimental): The treatment group will receive six hours follow-up and support weekly. The service will be provided by a dedicated Family Partner.
  Interventions: Behavioral: Family Partner
- Control group (No Intervention): The control group will receive default support from the child welfare services. The service will be "business as usual", provided by the local staff at the child welfare services.

INTERVENTIONS:
Behavioral: Family Partner — The Family Partner intervention is based on well-known elements for preventing child abuse and neglect, such as 1) high intensity intervention with home visitations, 2) coordination of services, 3) an ecological perspective, 4) parental guidance, and 5) an emphasis on a therapeutic relationship with parents to create trust, change and agency.
  Family Partners must have relevant professional background and education, such as social work, child welfare services and other health/welfare occupations. They must have a personal attitude for relation-based service delivery in a home-setting, a long work experience and in-depth knowledge of municipal welfare services.
  Each practitioner will follow five families. The estimated duration of the intervention is 12 months, but might go over longer stretches of time if it is considered beneficial for the families. The minimum duration of the intervention is 3 months.
  Arms: Experimental (Family Partner)

SUMMARY:
Prior to this pilot study, it is unclear whether comparing a manualized version of the Family Partner Model to standard practice in the Child Welfare Services would be feasible. Results will inform whether and how to design a fully powered randomized controlled trial to test the effects of a manualized version of the Family Partner Model on child maltreatment. The specific results of the pilot study will inform 1) randomization procedures, 2) data sources to be used, 3) sample size calculations, and 4) adaptations to the design and measures for a fully powered randomized controlled trial.

DETAILED DESCRIPTION:
The objective is to assess the adaptability and acceptability of the Family Partner Intervention, and the feasibility of a future randomised controlled trial. Our specific research questions are:

1. What is the adaptability, acceptability, and feasibility of the Family Partner intervention in a Norwegian municipal context?
2. What are the experiences and possible outcomes of the Family Partner intervention?
3. Is the trial design feasible for an RCT expansion?

The investigators will pilot a parallel randomized trial (RCT), allocated to two groups (treatment and control). Families that fit to the target group, will be invited to take part in the study. Each family which fit the inclusion criteria and consent to participate will be randomized with a 1:1 allocation to experimental and control groups. Each Family Partner can serve 5 families at a time, and the Family Partner will serve families from 6-18 months. As families complete the programme, new families will be recruited. Hence, the recruitment and randomization will be an ongoing process. Any changes to methods after pilot trial commencement will be reported along with study results.

In a future RCT, the objective is to evaluate the effectiveness of the Family Partner Intervention, i.e. whether introducing the intervention would improve the outcome of existing Child Welfare Services. Hence, the trial is a superiority trial, in which the Family Partner Intervention is hypothesized to be superior to existing service provision. The trial is designed according to an intention-to-treat principle, where all consented participants are included in the analyses, independent of their adherence to intervention.

ELIGIBILITY:
Inclusion criteria:

* parents are 18 years or older, and
* children are under 18 years, and
* families with complex challenges who are already involved in the Child Welfare Services, and
* children live under potentially harmful circumstances, and
* parents struggle in several areas, e.g. employment, poverty, drug misuse, mental health

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Acceptability | Acceptability at 12 months
  Intervention Rating Profile (IRP-15)

SECONDARY OUTCOMES:
Relationship between the Family Partner and the parents | Change from Baseline WAI at 3, 6, 9, 12, 15 and 18 months
  The Working Alliance Inventory (WAI)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Grete G Tøge, phd, Principal Investigator — associate professor; Eirin G Pedersen, phd, Principal Investigator — Senior Researcher
Locations (3):
- Norway (3):
  - Øvre Eiker kommune, Drammen
  - Larvik kommune, Larvik
  - Lillehammer kommune, Lillehammer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finne J, Toge AG, Wiggen KS, Ekre M, Malmberg-Heimonen I, Pontoppidan M, Dion J, Tommeras T, Pedersen E. Results from a randomized controlled pilot trial of a home-visiting intervention to reduce child maltreatment. Pilot Feasibility Stud. 2025 Jun 3;11(1):77. doi: 10.1186/s40814-025-01659-9. PMID 40462144
- [Derived] Pedersen E, Malmberg-Heimonen I, Finne J, Pontoppidan M, Dion J, Tommeras T, Toge AG. Family Partner: study protocol for a pilot randomised study of a home-visitation intervention in Norway. Scand J Public Health. 2024 Aug;52(6):761-768. doi: 10.1177/14034948231189773. Epub 2023 Aug 14. PMID 37574994